CLINICAL TRIAL: NCT00498966
Title: Phase II Study of Perifosine for Patients With Metastatic Carcinoma of the Kidney Who Have Progressed on a VEGF Receptor Inhibitor
Brief Title: Ph II Study of Perifosine for Patients With Carcinoma of the Kidney
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 231
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Kidney Cancer
Keywords: Kidney; perifosine; Progression on treatment with sunitinib or sorafenib
MeSH Terms: conditions — Kidney Neoplasms | interventions — perifosine

STUDY DESIGN:
Intervention Model Description: Two groups with regard to pre-treatment: patients in group A will have previously failed a VEGF receptor inhibitor but not an mTOR inhibitor, while patients in group B will have failed both a VEGF receptor inhibitor and an mTOR inhibitor.
  One treatment group: all patients will receive perifosine 100 mg qhs daily orally. Patients are to be instructed that perifosine is to be taken with food.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Patients in group A will have previously failed a VEGF receptor inhibitor but not an mTOR inhibitor.Intervention: Perifosine.
  Interventions: Drug: Perifosine
- Group B (Experimental): Patients in group B will have failed both a VEGF receptor inhibitor and an mTOR inhibitor. Intervention: Perifosine.
  Interventions: Drug: Perifosine

INTERVENTIONS:
Drug: Perifosine — Perifosine 100 mg PO Perifosine is supplied as a film-coated tablet containing 50 mg of active ingredient.
  Treatment will be administered on an outpatient basis in 28-day cycles. The patient dose for daily administration will be 100 mg qhs daily with food.
  Other Names: D-21266; KRX-0401

SUMMARY:
This is a Phase II study. Patients with kidney carcinoma will be considered in two groups. The goals of this study are:

* To measure clinical benefit defined as tumor response or progression-free survival for more than 12 weeks in patients with metastatic carcinoma of the kidney who have failed or have progressed on a VEGF receptor inhibitor
* To evaluate the safety of perifosine in patients with metastatic carcinoma of the kidney who have failed or have progressed on a VEGF receptor inhibitor

DETAILED DESCRIPTION:
This is a Phase II study. Patients with kidney carcinoma will be considered in two groups. Patients in group A will have previously failed a VEGF receptor inhibitor but not an mTOR inhibitor, while patients in group B will have failed both a VEGF receptor inhibitor and an mTOR inhibitor. Evaluation of each group will be performed separately. The goals of this study are:

1. To measure clinical benefit defined as an objective tumor response using RESIST or progression-free survival for more than 12 weeks in patients with metastatic carcinoma of the kidney who have failed or have progressed on a VEGF receptor inhibitor
2. To evaluate the safety of perifosine in patients with metastatic carcinoma of the kidney who have failed or have progressed on a VEGF receptor inhibitor.

Treatment Phase/duration of treatment: All patients will be treated with daily perifosine at 100 mg PO daily until tumor progression (by the RECIST criteria) or unacceptable toxicity. Once radiological disease progression has been documented by the treating physician, the patient will go off study. Patients are encouraged to have two measurements for confirmation of progression.

Follow-Up Phase: All patients will be followed-up for SAEs until at least 30 days after discontinuation of perifosine. All patients who are discontinued from perifosine for any reason other than disease progression will continue to have tumor assessments until the patient has documented disease progression or has begun other therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed metastatic RCC
* Patients must have documented progression on treatment with sunitinib or sorafenib. Prior therapy with bevacizumab and/or cytokines (i.e., IL-2, interferon) is permitted. Prior vaccine therapy in the adjuvant setting is also permitted. Patients can have failed therapy with ONE prior mTOR inhibitor.
* Patients must have at least one measurable lesion on computer tomography (CT) Scan or magnetic resonance imaging (MRI) using Modified RECIST criteria.
* Patients must have normal organ and marrow function, unless in the opinion of the treating investigator, the abnormality is related to tumor, and the study chairman agree the abnormality is unlikely to affect the safety of perifosine use. Normal organ and marrow function is described below:

  * ANC >= 1.5 x 109/L
  * Platelets >= 75,000/ mm3
  * HCT >= 28% (with or without growth factor support)
  * Creatinine <= 3.0 mg/dl
  * Total bilirubin <= 1.5 x upper limit of normal
  * Transaminase <= 2.5 x upper limit of normal
* ECOG performance status of 0 or 1
* Patients with CNS metastases must be clinically stable for at least 2 months following treatment with radiation therapy, surgery, or both; and be off corticosteroids and anti-seizure medication.
* Patients with a life expectancy ≥6 months
* Age ≥18 years old
* Patients who give a written informed consent obtained according to local guidelines
* Women of childbearing potential must have had a negative serum or urine pregnancy test 72 hours prior to the administration of the first study treatment.

Exclusion Criteria:

* Patients who have not recovered (<= grade 1) from adverse events from prior therapy (excluding alopecia).
* Patients currently receiving sorafenib or sunitinib who have received either of these within 2 weeks prior to study entry.
* Patients may have had prior sorafenib OR sunitinib BUT cannot have been treated with both VEGF receptor inhibitors.
* Patients with a known hypersensitivity to perifosine or its excipients.
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods.
* Patients who are using other investigational agents or who had received investigational drugs <= 4 weeks prior to study entry.
* Patients unwilling to or unable to comply with the protocol.
* Patients who have a history of another primary malignancy <= 5 years with the exceptions of non melanomatous skin cancer and carcinoma in situ of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-07; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Objective tumor response using RESIST OR progression-free survival | 12 weeks
  Clinical benefit, defined as either an objective response by RECIST or PFS >12 weeks, is a primary endpoint of the study. The clinical benefit rate together with its two-sided exact binomial 95% confidence interval will be reported.

SECONDARY OUTCOMES:
Evaluate the safety of perifosine in patients with metastatic carcinoma of the kidney | 12 weeks
  Safety endpoints include: incidence of adverse events, serious adverse events, change in vital signs and change in laboratory results (hematology, blood chemistry, urinalysis).

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Vogelzang, MD, Study Chair — Nevada Cancer Institute
Locations (3):
- United States (3):
  - Investigative Site, Louisville, Kentucky
  - Investigative Site, Morristown, New Jersey
  - Investigative Site, Armonk, New York

REFERENCES:
- [Result] Journal of Clinical Oncology, 2009 ASCO Annual Meeting Proceedings (Post-Meeting Edition). Vol 27, No 15S (May 20 Supplement), 2009: 5101